CLINICAL TRIAL: NCT02206997
Title: Evaluation of a Patient Warming Concept Following the New German Speaking S3 Guideline for Prevention of Intraoperative Hypothermia With Respect to Incidence and Complications of Perioperative Hypothermia
Brief Title: Evaluation of a Patient Warming Concept Following the German S3 Guideline for Prevention of Intraoperative Hypothermia
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, PD Dr. Jan Hoecker, MD, University Hospital Schleswig-Holstein
Other Study IDs: THER-GUIDE-EVA
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Hypothermia; Hypothermia, Accidental
Keywords: perioperative hypothermia; prewarming; treatment guideline
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Passive Insulation standard treatment: no active warming before start of anesthesia and no active warming at PACU
- Active prewarming treatment: active warming before start of anesthesia and active warming at PACU following recommendations of S3-guideline

SUMMARY:
The aim of the study is to evaluate a patient prewarming concept following the recommendations of the S3-guideline "Prevention of perioperative hypothermia" with respect to incidence and complications of perioperative hypothermia. The study hypothesis is that postoperative core temperature in adult patients after prewarming is significantly higher than in patients who were treated following actual standard protocol (passive insulation).

DETAILED DESCRIPTION:
The aim of the study is to evaluate a patient prewarming concept following the recommendations of the new german S3-guideline "Prevention of perioperative hypothermia" with respect to incidence and complications of perioperative hypothermia. Prewarming should enable the patients to preserve their core temperature for a longer period and to avoid perioperative hypothermia.The study hypothesis is that postoperative core temperature in adult patients after prewarming is significantly higher than in patients who were treated following the actual standard protocol (passive insulation).

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective general or orthopedic surgery with expected duration > 45 min
* American Society of Anesthesiologists physical status 1-3
* age > 17 years

Exclusion Criteria:

* emergency surgery
* patient's denial
* unexpected decrease of duration of anesthesia < 45 min
* preoperative body temperature > 38 °C

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of FEK Hospital Neumünster scheduled for elective surgery under defined conditions (see below)
Sampling Method: Non-Probability Sample
Enrollment: 485 (Actual)
Dates: Start 2014-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative hypothermia at admission to PACU | admission to PACU
  The incidence of postoperative hypothermia at admission to PACU should be evaluated by sublingual temperature measurement.

SECONDARY OUTCOMES:
Type and duration of surgery as influence factors for postoperative hypothermia at admission to PACU | admission to PACU
  Type and duration of surgery should be evaluated as influence factors for postoperative hypothermia at admission to PACU?

CONTACTS AND LOCATIONS:
Overall Officials: Jan H Hoecker, MD, Principal Investigator — University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Germany
Locations (1):
- FEK Hospital Neumünster, Neumünster, Schleswig-Holstein, Germany